CLINICAL TRIAL: NCT04881019
Title: Prediction of Glycemic Response Study (PROGRESS)
Brief Title: PRediction Of Glycemic RESponse Study
Acronym: PROGRESS
Status: Active, not recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: CareEvolution Healthcare Technology (Unknown); Tempus AI (Industry)
Responsible Party: Principal Investigator, Ed Ramos, Director, Digital Clinical Trials, Scripps Translational Science Institute
Other Study IDs: IRB-20-7635
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-12

CONDITIONS: Glycemic Response
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and stool for genetic and microbiome analyses, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Type 2 Diabetes: Individuals who have been diagnosed with Type 2 diabetes.
  Interventions: Device: Continuous glucose monitoring
- Non type 2 diabetes: Individuals who have not been diagnosed with Type 2 diabetes.
  Interventions: Device: Continuous glucose monitoring

INTERVENTIONS:
Device: Continuous glucose monitoring — Continuous monitoring of blood sugar over a 10-day period.
  Other Names: Dexcom G6

SUMMARY:
The purpose of PROGRESS is to engage and intensively monitor 1000 individuals' dietary intake, activity levels, and continuous glucose values over 10 days, link to clinical events out to 3-years, and use that data along with genomic, microbiome, electronic health record (EHR), and other biomarker data to develop a predictive model of individual glucose responses to nutrient intake in individuals with and without type 2 diabetes.

DETAILED DESCRIPTION:
Interested individuals will be directed to download the MyDataHelps™ (CareEvolution) mobile app to register and provide informed consent as well as prompt completion of surveys, share their electronic health record data and link the digital health technologies to be used in the study. Participants may be asked to schedule an initial virtual meeting (telephone or videoconference) with the research coordinator who will welcome and walk them through the study.

Once a participant has completed on-boarding, they will be asked to fill out a baseline health, lifestyle, and medical history surveys and, upon completion, invited to request a biosamples study kit to be delivered to their home. This biosamples kit will include:

* Salivary kit for genomics analysis
* Gut microbiome kit
* Home micro-puncture single-use blood collection

Additional study materials and devices include:

* A wrist-worn activity, heart rate and sleep monitor.
* A Dexcom 6 continuous glucose monitor (CGM) and application kit
* A standardized snack bar meal (2 per fasting days)

Participants will be asked to track various digital health measures including their continuous glucose as well as record their meals for a 10-day period. The data connections approved by the participants will continue in the following years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.

Exclusion Criteria:

* Type 1 diabetes mellitus
* Unable to participate in or comply with any of the testing modules asked during the study
* Currently pregnant
* Prior bariatric surgery
* Chemotherapy or radiation treatment for cancer in the past year
* Inflammatory bowel disease
* Known skin allergy to adhesives and nickel (or other contraindications to continuous glucose monitoring)
* Currently taking any oral steroids(these medications may impact glucose levels)
* Antibiotic use in the last 3 months prior to the start of the study or planned use during the duration of the study
* Non-dietary, supplemental probiotic use either daily or weekly
* Hospice care
* End stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be composed of 50% individuals with diagnosed T2D (using a validated algorithm) and 50% individuals without a formal diagnosis of T2D and who have a documented HgbA1C < 6.5 within the prior 2 years, matched to the T2D cohort based on age, gender, and BMI.
Sampling Method: Non-Probability Sample
Enrollment: 1070 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gylcemic response profiles | 10-days
  Distinguish differences in individual glycemic response characteristics as measured by the continuous glucose monitor (mg/dl) and macronutrients (carbohydrates, fats, and proteins) in participants with (n = 500) and without type 2 diabetes (n = 500) matched for age, sex, BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Ramos, PhD, Principal Investigator — Scripps Research
Locations (1):
- Scripps Research Translational Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided